CLINICAL TRIAL: NCT06716970
Title: A Multicenter, Randomized, Double-blind, and Active-controlled Parallel Study to Evaluate the Efficacy and Safety of QR12000 Compound Tablets and Sacubitril/valsartan Tablets in Patients with Moderate to Severe Essential Hypertension
Brief Title: QR12000 Compound Tablets in Patients with Moderate to Severe Essential Hypertension
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QR12000-GXY-3-01
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — sacubitril; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- QR12000 75mg (Experimental): Participants will be treated with one tablet of QR12000 75mg, one tablet of QR12000 150mg placebo and one tablet of Sacubitril/valsartan 200 mg placebo once daily for up to 8 weeks. Participants continue with one tablet of QR12000 150mg once daily for 44 weeks during TOP observation period.
  Interventions: Drug: QR12000 75mg; Drug: QR12000 150mg placebo; Drug: Sacubitril/valsartan 200mg placebo
- QR12000 150mg (Experimental): Participants will be treated with one tablet of QR12000 150mg, one tablet of QR12000 75mg placebo and one tablet of Sacubitril/valsartan 200 mg placebo once daily for up to 8 weeks. Participants continue with one tablet of QR12000 150mg once daily for 44 weeks during TOP observation period.
  Interventions: Drug: QR12000 75mg placebo; Drug: QR12000 150mg; Drug: Sacubitril/valsartan 200mg placebo
- Sacubitril/valsartan 200 mg (Active Comparator): Participants will be treated with one tablet of Sacubitril/valsartan 200 mg, one tablet of QR12000 75mg placebo and one tablet of QR12000 150mg placebo once daily for up to 8 weeks. Participants continue with one tablet of QR12000 150mg once daily for 44 weeks during TOP observation period.
  Interventions: Drug: QR12000 75mg placebo; Drug: QR12000 150mg placebo; Drug: Sacubitril/valsartan 200mg

INTERVENTIONS:
Drug: QR12000 75mg — QR12000 75mg QD
  Arms: QR12000 75mg
Drug: QR12000 75mg placebo — Matching placebo of QR12000 75mg QD
  Arms: QR12000 150mg; Sacubitril/valsartan 200 mg
Drug: QR12000 150mg — QR12000 150mg QD
  Arms: QR12000 150mg
Drug: QR12000 150mg placebo — Matching placebo of QR12000 150mg QD
  Arms: QR12000 75mg; Sacubitril/valsartan 200 mg
Drug: Sacubitril/valsartan 200mg — Sacubitril/valsartan 200mg QD
  Arms: Sacubitril/valsartan 200 mg
Drug: Sacubitril/valsartan 200mg placebo — Matching placebo of Sacubitril/valsartan 200mg QD
  Arms: QR12000 150mg; QR12000 75mg

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of QR12000 75mg, QR12000 150mg and Sacubitril/valsartan 200mg in patients with moderate to severe essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who can understand and are willing to complying with protocol requirement and sign the informed consent form.
2. Man or woman aged 18 years to 75 years (inclusive), with BMI≤30 kg/m2.
3. Patients with moderate to severe hypertension. Untreated patients must have an msSBP ≥ 160 mmHg and < 190 mmHg at the screening and randomization visit; Treated patients must have an msSBP≥150 mmHg and <180 mmHg or msSBP≥140 mmHg and <170 mmHg at the screening visit based on numbers of antihypertensive and msSBP≥160 mmHg <190 mmHg at the randomization visit; Patients must have an absolute difference of ≤20 mmHg in msSBP between randomization visit and the immediately preceding visit.
4. Subjects who agree to use adequate contraception from 2 weeks prior to screening to 1 month after last dose.

Exclusion Criteria:

1. History or evidence of a secondary form of hypertension.
2. History of peripheral arterial occlusive disease and Raynaud's syndrome.
3. History of hyperthyroidism.
4. History of hypotension.
5. History of angioedema, drug-related or otherwise.
6. Suffered by severe cerebrovascular disease within 1 year prior to screening.
7. Suffered by severe heart disease within 1 year prior to screening
8. History of severe or malignant retinopathy.
9. History of aortic aneurysm or dissection, cardiac surgery, or percutaneous coronary intervention within 1 year prior to screening.
10. History of malignant tumor within 5 years prior to screening.
11. Poorly controlled diabetes prior to screening
12. History of severe autoimmune diseases.
13. History of severe mental disorder.
14. Clinically significant laboratory abnormalities.
15. History of allergy to the test drug, active control drug, or drugs similar to the test drug and positive control drug or related excipients.
16. Undergone gastrointestinal surgery that could significantly alter drug absorption, distribution, metabolism, and excretion, or with severe gastrointestinal diseases, dysphagia, or recurrent vomiting that causes difficulty in eating or taking medication.
17. Intolerance to the run-in period.
18. Poor medication compliance or other non-compliance during run-in period.
19. Participated in any interventional clinical trial within 3 months prior to screening, plan to participate in another clinical trial during the period of this trial, or plan to participate in another clinical trial within 1 month after the end of this trial.
20. History of alcohol abuse within 6 months prior to screening or evidence of drug abuse.
21. Not agree or unable to comply with the restrictions on concomitant treatment during the study.
22. Pregnancy test positive, lactating women, or women planning to become pregnant.
23. High-altitude workers or large motor vehicle drivers and other professionals engaged in hazardous mechanical operations.
24. Other conditions that by the investigator's discretion may interfere with efficacy or safety assessment of the study, or pose a great risk to the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) | Baseline and week 8
  The change in msSBP measured at Week 8 relative to baseline.

SECONDARY OUTCOMES:
Change From Baseline in Mean Sitting Diastolic BP (msDBP) | Baseline and week 8
  The change in msDBP measured at Week 8 relative to baseline.
Change From Baseline in Mean Ambulatory Systolic/Diastolic BP (maSBP/maDBP) | Baseline and week 8
  The change in maSBP/maDBP measured at Week 8 relative to baseline.
Change From Baseline in Daytime ( > 6am and ≤ 10 pm) or Nighttime (> 10 pm and ≤ 6 am) maSBP/maDBP | Baseline and week 8
  The change in Daytime or Nighttime maSBP/maDBP measured at Week 8 relative to baseline.
Percentage of Participants Achieving BP Control | Baseline and week 8
  BP control is defined as msSBP <140 mm Hg and msDBP <90 mm Hg.
Percentage of Participants Achieving BP Response | Baseline and week 8
  BP Response is defined as msSBP <140 mm Hg and/or a reduction of ≥20 mm Hg from Baseline and msDBP <90 mm Hg and/or a reduction of ≥10 mm Hg from Baseline.
Change From Baseline in msSBP/msDBP | Baseline, week 28 and week 52
  The change in msSBP/msDBP measured at Week 28 and Week 52 relative to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China